CLINICAL TRIAL: NCT05258981
Title: Exploring the Relationship Between Advanced Multimodal Brain MRI Phenotypes, Genes and Cognitive Outcome in Adults With CHD
Brief Title: The Relationship Between Brain MRI Phenotypes, Genes and Cognitive Outcome in CHD Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michelle Gurvitz, Associate Professor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P00039087
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain MRI (Other): Obtain Brain MRI in adults with congenital heart disease and age/sex matched controls
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Brain MRI

SUMMARY:
The main purpose of this proposal is to perform novel MRI analyses to determine the brain organizational changes associated with altered executive function and the modulating role of variants in neuroresilience and hypoxia response genes in adults with d-transposition of the great arteries (d-TGA).

DETAILED DESCRIPTION:
Aim 1 is structured to determine the relationship between sulcal patterns(measured by MRI) and executive function in adults with d-TGA and if this relationship is modified by (a) presence of neuroresilience gene ApoE ε2 or ε4 alleles, or (b) damaging variants in hypoxia response genes.

Aim 2 is designed to determine the relationship between structural connectivity using rich club (measured by MRI) and executive function in adults with d-TGA and if this relationship is modified by (a) presence of neuroresilience gene ApoE ε2 or ε4 alleles or (b) damaging variants in hypoxia response genes.

In Aim 3, the investigators will determine the relationship between functional connectivity using rich club (measured by MRI) and executive function in adults with d-TGA and if this relationship is modified by (a) presence of neuroresilience gene ApoE ε2or ε4 alleles or (b) damaging variants in hypoxia response genes.

ELIGIBILITY:
Inclusion Criteria:

* Persons who participated in the Boston circulatory arrest, pH and Hematocrit studies at Boston Childrens Hospital as children (n~300).
* Normally-developed age- and sex-matched young adults who are able to provide informed consent to undergo the MRI portion of the study and limited neuropsychological evaluation (IQ assessment as well as neuropsychological tests for which normative references are not available).

Exclusion Criteria:

* For controls - inability to complete the MRI (implanted metal, claustrophobia, personal history of mental illness, brain injury, prior brain intervention).
* Intellectual impairment precluding completion of the study questionnaires independently
* Unable to speak and read English fluently

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Delis-Kaplan Executive Function Scale (D-KEFS) composite score; | Baseline
  measure of executive function

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared with other researchers upon request and approval of the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available 5 years after study completion
Access Criteria: Researchers will need to request the data and have approval of the study PI